CLINICAL TRIAL: NCT06424691
Title: Infant Restore: Investigating the Efficacy of a Microbiome Analysis, Education, and Recommendation Program in Improving Infant Gut Health
Brief Title: Infant Restore: Efficacy of Microbiome Analysis and Education
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seeding, Inc DBA Tiny Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IR-001
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Microbiota; Eczema; Microbiome; Gut Microbiome
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will receive comprehensive support to improve their infant's gut health over six months.
  Interventions: Dietary Supplement: Tailored Recommendations; Behavioral: Consult Call; Behavioral: Email Series
- Control (No Intervention): Participants in the control arm will serve as a comparison group and will not receive the intervention during the study period.

INTERVENTIONS:
Dietary Supplement: Tailored Recommendations — Based on the microbiome analysis, participants will receive personalized action plans. These plans include dietary, lifestyle, and supplemental suggestions to improve their infant's gut health.
  Arms: Intervention
Behavioral: Consult Call — Participants will have seven consult calls with a Gut Health Coach over the course of the study. These calls will provide guidance on the gut health reports, action plans, and any questions or concerns parents may have.
  Arms: Intervention
Behavioral: Email Series — Parents will receive a series of educational emails covering topics such as the importance of gut health, breastfeeding benefits, the impact of C-section delivery on the microbiome, and tips for introducing solid foods.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn if a microbiome analysis, education, and recommendation program can improve gut health, reduce future health risks, and empower parents in their children's health in infants aged 0-3 months delivered via Cesarean section. The main questions it aims to answer are: Will the intervention increase bacteria considered beneficial, decrease the C- section microbiome signatures, promote a reduction in opportunistic pathogens, and improved functional potential for HMO digestion and SCFA production Will the intervention decrease microbiome signatures associated with atopic march conditions.

Researchers will compare participants in the intervention arm, who will receive microbiome reports, personalized action plans, and educational materials, to participants in the control arm, who will receive microbiome results and educational materials after the study's completion, to see if the intervention leads to improved gut health and reduced risk of health conditions.

Participants will:

* Provide two microbiome stool samples three months apart.
* Receive detailed infant gut health reports via the Tiny Health app.
* Receive personalized action plans tailored to their infant's gut health needs.
* Engage in gut health coaching sessions with a microbiome expert.
* Receive an educational email series on infant gut health.
* Complete a series of surveys/questionnaires on health history, symptoms, and diet.

This study seeks to demonstrate that targeted microbiome interventions can significantly improve early infant gut health, leading to potential long-term health benefits. These benefits may include reduced healthcare costs by lowering the incidence of related chronic conditions. By establishing a foundation for mitigating these conditions, the intervention could consequently result in fewer doctor visits, reduced need for medications, and a lower incidence of hospitalizations over the first 3-4 years of the infant's life.

ELIGIBILITY:
Inclusion Criteria:

* Infants are qualified for this study if they are 0 to 3 months of age at time of enrollment.
* Infant was delivered via Cesarean delivery (C-section).

Exclusion Criteria:

* Infants cannot have been given probiotic supplements in their life at recruitment. This includes probiotic powder or supplements or formula with probiotic addition or multivitamin with probiotic addition.
* Twin and multiple birth infants are not accepted in this study.
* Infants must be full term or no less than 36-weeks gestation at delivery.
* Infants must be residents of the United States with US postal service.
* Infants cannot have the following existing health conditions:

  * Pre-existing gut conditions (Hirschsprung disease, eosinophilic gastrointestinal disorders (EGID) such as eosinophilic esophagitis (EoE), necrotizing enterocolitis (NEC), short bowel syndrome (SBS))
  * Immune or auto-immune conditions (severe combined immunodeficiency (SCID), human immunodeficiency virus (HIV)), excluding eczema and rashes
  * Congenital conditions (cleft lip or cleft palate, congenital heart disease, cerebral palsy, fragile X syndrome, down syndrome, spina bifida, cystic fibrosis, phenylketonuria (PKU), congenital hypothyroidism (CHT), galactosaemia)
  * Blood disorders (sickle cell disease, thalassemia, hemophilia)
* Infants are excluded if they or any of their immediate family members have received results from an at-home microbiome stool test in the past. This does not include clinical workup such as culture or pathogen testing.

Ages: 0 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-04-14 (Estimated); Study Completion 2025-04-14 (Estimated)

PRIMARY OUTCOMES:
Microbiota composition | 6 months
  Assess changes in beneficial bacteria (Bifidobacterium) and C-section microbiome signatures. Detect levels of opportunistic pathogens, and changes in functional potential for HMO digestion and SCFA production.

SECONDARY OUTCOMES:
C-section signature | 6 months
  Detect signature shifts from a C-section signature to a vaginally born signature
Atopic march signature | 6 months
  Compare atopic march signatures of intervention arm versus control subjects

OTHER OUTCOMES:
Educational | 6 months
  Asses parental understanding and engagement in gut health.
Gut reacted symptoms | 6 months
  Measure changes in newborn symptoms known to be influenced by gut microbiome e.g. colic, GI upset, sleep issues, eczema.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Sukhum, PhD, Principal Investigator — Seeding INC
Locations (1):
- Seeding INC, Fredericksburg, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galazzo G, van Best N, Bervoets L, Dapaah IO, Savelkoul PH, Hornef MW; GI-MDH consortium; Lau S, Hamelmann E, Penders J. Development of the Microbiota and Associations With Birth Mode, Diet, and Atopic Disorders in a Longitudinal Analysis of Stool Samples, Collected From Infancy Through Early Childhood. Gastroenterology. 2020 May;158(6):1584-1596. doi: 10.1053/j.gastro.2020.01.024. Epub 2020 Jan 18. PMID 31958431
- [Background] Shao Y, Forster SC, Tsaliki E, Vervier K, Strang A, Simpson N, Kumar N, Stares MD, Rodger A, Brocklehurst P, Field N, Lawley TD. Stunted microbiota and opportunistic pathogen colonization in caesarean-section birth. Nature. 2019 Oct;574(7776):117-121. doi: 10.1038/s41586-019-1560-1. Epub 2019 Sep 18. PMID 31534227
- [Background] O'Neill I, Schofield Z, Hall LJ. Exploring the role of the microbiota member Bifidobacterium in modulating immune-linked diseases. Emerg Top Life Sci. 2017 Nov 30;1(4):333-349. doi: 10.1042/ETLS20170058. PMID 33525778
- [Background] Roswall J, Olsson LM, Kovatcheva-Datchary P, Nilsson S, Tremaroli V, Simon MC, Kiilerich P, Akrami R, Kramer M, Uhlen M, Gummesson A, Kristiansen K, Dahlgren J, Backhed F. Developmental trajectory of the healthy human gut microbiota during the first 5 years of life. Cell Host Microbe. 2021 May 12;29(5):765-776.e3. doi: 10.1016/j.chom.2021.02.021. Epub 2021 Mar 31. PMID 33794185
- [Result] Vandenplas Y, De Greef E, Veereman G. Prebiotics in infant formula. Gut Microbes. 2014;5(6):681-7. doi: 10.4161/19490976.2014.972237. PMID 25535999
- [Derived] Nieto PA, Nakama C, Trachsel J, Goad D, Soderborg TK, Tan DS, Orlandi A, Yuan Q, Song E, Mueller NT, Mars RA, Hoy CS, Sukhum KV. Improving immune-related health outcomes post-cesarean birth with a gut microbiome-based program: A randomized controlled trial. Pediatr Allergy Immunol. 2025 Sep;36(9):e70182. doi: 10.1111/pai.70182. PMID 40898384